CLINICAL TRIAL: NCT05760911
Title: A Multi-center Clinical Study on the Myopia Prevention by Monitoring and Motivating Outdoor Activities With Smartwatches
Brief Title: Myopia Prevention Through Monitoring and Motivating Outdoor Activities With Smartwatches
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: kjb-wb-v1.1-20220507
Record Dates: First submitted 2023-02-15; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Myopia, Progressive
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outdoor activities motivating group (Experimental): Wear a smartwatch and receive Mini Program reminders and encouragement for outdoor activities. The required outdoor time is at least 2 hours from Monday to Friday and more than 2 hours on weekends.
  Interventions: Behavioral: Outdoor activities motivation with smartwatches
- Outdoor activities monitoring group (No Intervention): Outdoor activities are monitored with smartwatches.

INTERVENTIONS:
Behavioral: Outdoor activities motivation with smartwatches — Wearing a smartwatch and receiving outdoor activity reminders and encouragement through a mini-program. The required outdoor time is at least 2 hours from Monday to Friday, and more than 2 hours on weekends.
  Arms: Outdoor activities motivating group

SUMMARY:
The goal of this multi-center, randomized, parallel-controlled clinical trial is to evaluate the effectiveness of outdoor activities monitoring and motivating by smartwatches to prevent myopia progression in children. The main question it aims to answer are:

1. To evaluate the two-year change of spherical equivalent progression.
2. To evaluate the change in axial length, the incidence of myopia, the time of outdoor activity, the choroid thickness, and blood flow through the two-year intervention.

Participants will wear smartwatches and receive Mini Program outdoor activity reminders and motivations. The required outdoor activity time is 2 hours from Monday to Friday and more than 2 hours on weekends. The control group will only wear smartwatches for monitoring. Researchers will compare the control group and the intervention group to see if outdoor activities can protect myopia or not.

ELIGIBILITY:
Inclusion Criteria:

1. Gender is not limited;
2. Age: 4 ~ 9 years old;
3. Spherical equivalent: -0.5D < SE < 2.5D;
4. Be able to follow up for at least 2 years;
5. Be able to wear a smartwatch on a daily basis as required;
6. Parents or guardians sign an informed consent form;
7. Children over 6 years old need oral consent to participate.

Exclusion Criteria:

1. Anisometropia > 1.50D;
2. Using other interventions for controlling myopia including atropine, rigid orthokeratology lenses, bifocal lenses or progressive lenses, red light, acupuncture, etc.;
3. Strabismus and/or amblyopia;
4. Previous history of eye surgery (including strabismus correction);
5. Ocular or systemic diseases that may be related to the development of myopia or myopia: such as Marfan syndrome, neonatal retinopathy, diabetes, etc.;
6. Other circumstances that the investigator judges inappropriate to participate in the trial.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The change of spherical equivalent | Two years
  The mean change of spherical equivalent after cycloplegia was calculated during the study.

SECONDARY OUTCOMES:
The change of axial length | Two years
  The mean change of axial length by IOL Master was calculated during the study.

IPD SHARING:
Plan to Share IPD: No